CLINICAL TRIAL: NCT07148674
Title: Efficacy of Positive Expiratory Pressure on Acute Mountain Sickness, a Pilot Crossover Trial at 6000 Meters
Brief Title: Efficacy of Positive Expiratory Pressure on Acute Mountain Sickness
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BiALP - Alpine, Disaster and Wilderness Medicine (Other)
Collaborators: Società Italiana Medicina degli Ambienti Estremi (Unknown)
Responsible Party: Principal Investigator, Paolo Rodi, MD, MScMD, principal investigator, BiALP - Alpine, Disaster and Wilderness Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6962
Record Dates: First submitted 2025-08-06; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Acute Mountain Sickness (AMS)
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Pilot trial of positive expiratory pressure for acute mountain sickness.
  1 single arm with 3 phases:
  * 1: Baseline Breathing (No PEP) Participants breathe normally without any device for 10 minutes in supine position, serving as control.
  * 2: Positive Expiratory Pressure (PEP) Breathing Participants breathe through a face mask with a mechanical PEP device set at 10 cmH₂O expiratory pressure for 10 minutes supine. Inspiration is unrestricted; expiration occurs against resistance to improve oxygenation and reduce AMS symptoms.
  * 3: Post-PEP Breathing (No PEP) After PEP, participants breathe normally for 10 minutes supine.
  Each phase is consecutive at altitudes 4,300 m, 5,560 m, and 6,000 m
  Interventions: Device: Positive Expiratory Pressure (10cmH2O) in hypobaric hypoxia

INTERVENTIONS:
Device: Positive Expiratory Pressure (10cmH2O) in hypobaric hypoxia — The intervention under investigation will be the application of positive expiratory pressure (PEP) at 10 cmH₂O using an Ambu mask. The mask will allow participants to inspire freely while generating a controlled expiratory pressure. The PEP device is a non-pharmacological medical device whose uses in both hospital and pre-hospital settings are part of everyday medical practice.

SUMMARY:
This pilot study aims to evaluate the efficacy of positive expiratory pressure (PEP) therapy at 10 cmH₂O in improving peripheral oxygen saturation (SpO₂) and mitigating symptoms of acute mountain sickness (AMS) in healthy individuals exposed to extreme altitude conditions.

Three male participants will be monitored during an ascent of Mount Aconcagua, Argentina, at elevations of 4,300 m, 5,560 m, and 6,000 m above sea level. The study involves three sequential phases of 10 minutes each: baseline breathing without PEP, breathing with PEP applied via a mechanical face mask, and post-PEP breathing.

Primary outcomes include changes in SpO₂ and Lake Louise Score (LLS) to assess AMS severity. Findings will provide preliminary data on the potential role of PEP as a non-pharmacological intervention in high-altitude medicine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers without ongoing medical conditions
* Over 18 years of age
* Volunteers with the physical and technical skills necessary to undertake a mountaineering expedition on Mount Aconcagua, Argentina, and with previous experience at extreme altitudes

Exclusion Criteria:

* Subjects with any ongoing medical conditions
* Under 18 years of age
* Subjects without previous mountaineering experience at extreme altitudes and without adequate physical and technical preparation necessary to undertake a mountaineering expedition on Mount Aconcagua, Argentina

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-09-05 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Peripheral Oxygen Saturation (SpO2) | During the 3 weeks of expedition on Mount Aconcagua, after arrival of participants at 4300masl, 5560masl and 6000 masl.

SECONDARY OUTCOMES:
Lake Louise Score | During the 3 weeks of expedition on Mount Aconcagua, after arrival of participants at 4300masl, 5560masl and 6000 masl.
  The Lake Louise Score (LLS) is a standardized tool to diagnose Acute Mountain Sickness (AMS). It combines self-reported symptoms (headache, gastrointestinal upset, fatigue/weakness, dizziness/lightheadedness) rated from 0 (none) to 3 (severe). AMS is diagnosed when headache is present plus at least one other symptom, with a total score ≥3. Higher scores reflect greater symptom severity: 3-5 mild AMS, 6-9 moderate, ≥10 severe. The LLS is used in research and expeditions to quantify altitude illness and monitor response to acclimatization or treatment.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mellor A. Research at high altitudes. J R Army Med Corps. 2011 Mar;157(1):5-7. doi: 10.1136/jramc-157-01-01. PMID 21465903
- [Background] Wu J, Wu Y, Wang L, Ye H, Lu J, Li Y. Challenges and Advances in Rechargeable Batteries for Extreme-Condition Applications. Adv Mater. 2024 Jan;36(4):e2308193. doi: 10.1002/adma.202308193. Epub 2023 Nov 28. PMID 37847882
- [Background] Nespoulet H, Rupp T, Bachasson D, Tamisier R, Wuyam B, Levy P, Verges S. Positive expiratory pressure improves oxygenation in healthy subjects exposed to hypoxia. PLoS One. 2013 Dec 23;8(12):e85219. doi: 10.1371/journal.pone.0085219. eCollection 2013. PMID 24376872
- [Background] Johnson PL, Johnson CC, Poudyal P, Regmi N, Walmsley MA, Basnyat B. Continuous positive airway pressure treatment for acute mountain sickness at 4240 m in the Nepal Himalaya. High Alt Med Biol. 2013 Sep;14(3):230-3. doi: 10.1089/ham.2013.1015. PMID 24067184
- [Background] Rupp T, Saugy JJ, Bourdillon N, Verges S, Millet GP. Positive expiratory pressure improves arterial and cerebral oxygenation in acute normobaric and hypobaric hypoxia. Am J Physiol Regul Integr Comp Physiol. 2019 Nov 1;317(5):R754-R762. doi: 10.1152/ajpregu.00025.2019. Epub 2019 Sep 18. PMID 31530174
- [Background] Rupp T, Maufrais C, Walther G, Esteve F, Macdonald JH, Bouzat P, Verges S. MEDEX 2015: Prophylactic Effects of Positive Expiratory Pressure in Trekkers at Very High Altitude. Front Physiol. 2021 Sep 21;12:710622. doi: 10.3389/fphys.2021.710622. eCollection 2021. PMID 34621182
- [Background] Fagevik Olsen M, Lannefors L, Westerdahl E. Positive expiratory pressure - Common clinical applications and physiological effects. Respir Med. 2015 Mar;109(3):297-307. doi: 10.1016/j.rmed.2014.11.003. Epub 2014 Nov 12. PMID 25573419
- [Background] Gabry AL, Ledoux X, Mozziconacci M, Martin C. High-altitude pulmonary edema at moderate altitude (< 2,400 m; 7,870 feet): a series of 52 patients. Chest. 2003 Jan;123(1):49-53. doi: 10.1378/chest.123.1.49. PMID 12527602
- [Background] Agostoni P, Caldara G, Bussotti M, Revera M, Valentini M, Gregorini F, Faini A, Lombardi C, Bilo G, Giuliano A, Veglia F, Savia G, Modesti PA, Mancia G, Parati G; HIGHCARE Investigators. Continuous positive airway pressure increases haemoglobin O2 saturation after acute but not prolonged altitude exposure. Eur Heart J. 2010 Feb;31(4):457-63. doi: 10.1093/eurheartj/ehp472. Epub 2009 Nov 10. PMID 19903683
- [Background] Wang C, Wang X, Chi C, Guo L, Guo L, Zhao N, Wang W, Pi X, Sun B, Lian A, Shi J, Li E. Lung ventilation strategies for acute respiratory distress syndrome: a systematic review and network meta-analysis. Sci Rep. 2016 Mar 9;6:22855. doi: 10.1038/srep22855. PMID 26955891
- [Background] Roach RC, Hackett PH, Oelz O, Bartsch P, Luks AM, MacInnis MJ, Baillie JK; Lake Louise AMS Score Consensus Committee. The 2018 Lake Louise Acute Mountain Sickness Score. High Alt Med Biol. 2018 Mar;19(1):4-6. doi: 10.1089/ham.2017.0164. Epub 2018 Mar 13. PMID 29583031
- [Background] Luks AM, Beidleman BA, Freer L, Grissom CK, Keyes LE, McIntosh SE, Rodway GW, Schoene RB, Zafren K, Hackett PH. Wilderness Medical Society Clinical Practice Guidelines for the Prevention, Diagnosis, and Treatment of Acute Altitude Illness: 2024 Update. Wilderness Environ Med. 2024 Mar;35(1_suppl):2S-19S. doi: 10.1016/j.wem.2023.05.013. Epub 2023 Dec 27. PMID 37833187
- [Background] Woods P, Alcock J. High-altitude pulmonary edema. Evol Med Public Health. 2021 Jan 6;9(1):118-119. doi: 10.1093/emph/eoaa052. eCollection 2021. PMID 33732460
- [Background] Hackett PH, Rennie D, Levine HD. The incidence, importance, and prophylaxis of acute mountain sickness. Lancet. 1976 Nov 27;2(7996):1149-55. doi: 10.1016/s0140-6736(76)91677-9. PMID 62991
- [Background] Netzer N, Strohl K, Faulhaber M, Gatterer H, Burtscher M. Hypoxia-related altitude illnesses. J Travel Med. 2013 Jul-Aug;20(4):247-55. doi: 10.1111/jtm.12017. Epub 2013 Mar 11. PMID 23809076
- See also: Theoretical underpinning — https://pubmed.ncbi.nlm.nih.gov/34621182/
- See also: Theoretical underpinning — https://pubmed.ncbi.nlm.nih.gov/31530174/